CLINICAL TRIAL: NCT02971280
Title: Influence of Heavy Metals Exposure on in Vitro Fertilization (IVF) Outcome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Shahar Kol MD, Director IVF Unit, principal investigator, Assistant clinical Professor, Rambam Health Care Campus
Other Study IDs: 0008-16-RMB
Record Dates: First submitted 2016-11-14; First posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Fertilization in Vitro

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Exposure to heavy metals may interfere with basic cellular functions, including DNA synthesis.

The aim of the study is to correlate heavy metals concentration in body fluids of reproductive importance and IVF outcome.

DETAILED DESCRIPTION:
Concentration of heavy metals will be measured in blood, urine, semen fluid and follicular fluid of IVF patients.

Study group: poor prognosis patients: repeated IVF failure, implantation failure, poor ovarian response, low sperm quality (according to WHO criteria) Control group: Good prognosis patients. Normal sperm count. Heavy metals concentrations will be measured using atomic absorption spectrometer, and will be correlated with IVF outcomes: number of mature oocytes obtained, fertilizations, embryos quality, and reproductive outcome post embryo transfer.

ELIGIBILITY:
Inclusion Criteria

* Age of female patients: <=39
* Age of male patients: 18-50

Exclusion Criteria:

* Smoking
* Alcohol/drug abuse
* Long-term/chronic medications
* Severe health/mental problems
* Dental or other transplants
* Fragile X mutations
* Fertility preservation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: IVF patients (women and men)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Live birth rate ("take-home baby") | 9 months from embryo transfer
  IVF cycle resulting in pregnancy that ends in a live birth.

SECONDARY OUTCOMES:
Clinical pregnancy rate | 1 month from embryo transfer
  Gestational sac(s) seen by ultrasound 1 month after embryo transfer.

IPD SHARING:
Plan to Share IPD: No
Data will be published in scientific journal. Individual researchers will have access to source data anonymously.